CLINICAL TRIAL: NCT03522649
Title: A Phase III, Randomized, Open-Label Clinical Study of Napabucasin (GB201) in Combination With FOLFIRI Versus Napabucasin in Adult Patients With Previously Treated Metastatic Colorectal Cancer (CRC)
Brief Title: A Phase III Clinical Study of Napabucasin (GB201) Plus FOLFIRI in Adult Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 1Globe Health Institute LLC (Industry)
Responsible Party: Sponsor
Organization: 1Globe Biomedical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEMNESS-CRC
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Previously Treated Metastatic Colorectal Cancer
Keywords: CRC
MeSH Terms: interventions — napabucasin; Fluorouracil; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Napabucasin plus FOLFIRI (Experimental): Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 8~12 hours. For patients who have failed bevacizumab with irinotecan-based chemotherapies, bevacizumab may be administered with FOLFIRI. FOLFIRI infusion will start at least 2 hours following the first daily dose of napabucasin and will be administered every 2 weeks, starting on C1D1. If bevacizumab is added to FOLFIRI, bevacizumab infusion should start at least 2 hours following the first daily dose of napabucasin and will be administered every 2 weeks. Irinotecan/leucovorin infusion will follow bevacizumab infusion. 5-FU 400 mg/ m^2 bolus will be administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/ m^2/day continuous infusion. For patients who could not tolerate FOLFIRI at the full dose previously, FOLFIRI should be started at the same dose level the patient tolerated FOLFIRI previously.
  Interventions: Drug: Napabucasin; Drug: Fluorouracil; Drug: Leucovorin; Drug: Irinotecan
- Napabucasin (Other): Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 8~12 hours.
  Interventions: Drug: Napabucasin

INTERVENTIONS:
Drug: Napabucasin — Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 8~12 hours.
  Other Names: GB201
Drug: Fluorouracil — Fluorouracil 400 mg/m^2 bolus will be administered intravenously immediately following irinotecan/leucovorin infusion, followed by Fluorouracil 1200 mg/m^2/day (total 2400 mg/m^2) continuous infusion.
  Other Names: 5-FU; Benda-5 FU
  Arms: Napabucasin plus FOLFIRI
Drug: Leucovorin — Irinotecan 180 mg/m^2 followed by or concurrent with leucovorin 400 mg/m^2 will be administered intravenously, over approximately 90 minutes and 2 hours, respectively.
  Other Names: Folinic Acid
  Arms: Napabucasin plus FOLFIRI
Drug: Irinotecan — Irinotecan 180 mg/m^2 followed by or concurrent with leucovorin 400 mg/m^2 will be administered intravenously, over approximately 90 minutes and 2 hours, respectively.
  Other Names: Irinotecan Aurobindo
  Arms: Napabucasin plus FOLFIRI

SUMMARY:
This is a randomized, open-label, multi-center, phase III study of Napabucasin plus bi-weekly FOLFIRI (Arm 1) vs. Napabucasin (Arm 2) for adult patients with metastatic CRC who have failed standard chemotherapy regimens. For patients who have failed bevacizumab with irinotecan-based chemotherapies (treatment failure is defined as radiologic progression of disease during or within 3 months following the last dose), bevacizumab maybe administered in combination with FOLFIRI to patients randomized to Arm 1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum that is metastatic (Stage IV)
* Progression during or within 3 months following the last administration of standard chemotherapy based regimens containing a fluoropyrimidine, irinotecan and oxaliplatin. Patients treated with oxaliplatin or irinotecan in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy
* Patients who are candidates for and have access to anti-VEGF therapy (i.e. bevacizumab and regorafenib) and anti-EGFR therapy (i.e. cetuximab and panitumumab) and/or TAS-102 must have received appropriate therapy.
* Patients with measurable or non measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of </= 1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Anti-cancer chemotherapy, biologic therapy or any other systemic therapy if administered prior to the first planned dose of study medication within period of time equivalent to the usual cycle length of the regimen. An exception is made for oral fluoropyrimidines (e.g. capecitabine, S-1), where a minimum of 10 days since last dose must be observed prior to the first planned dose of protocol treatment.
* Major surgery within 4 weeks prior to randomization.
* Any known brain or leptomeningeal metastases are excluded, even if treated.
* Known hypersensitivity to 5-FU/LV or patients who as a result of toxicity had to reduce or stop 5-FU infusion at the dose of 900 mg/m^2/day (total 1800 mg/m^2/day).
* Known hypersensitivity to irinotecan or patients who as a result of toxicity had to reduce or stop irinotecan infusion at the dose of 120 mg/m^2.
* Known history of human immunodeficiency virus (HIV) infection. Known chronic hepatitis B or C active infection.
* Known microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR).
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Patients with QTc interval > 470 millisecond.
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 43 months
  To assess the effect of Napabucasin plus biweekly FOLFIRI versus Napabucasin on the Overall Survival of patients with previously treated metastatic colorectal cancer.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 43 months
  Defined as the time from randomization to the first objective documentation of disease progression or death due to any cause.
Objective response rate (ORR) | 43 months
  Defined as the proportion of patients with a documented complete response or partial response (CR + PR) based on RECIST 1.1.
Disease control rate (DCR) | 43 months
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Number of Patients with Adverse Events | 43 months
  All patients who have received at least one dose of Napabucasin will be included in the safety analysis according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.0. The incidence of adverse events will be summarized by type of adverse event and severity.
Quality of Life (QoL) | 43 months
  QoL will be measured using the European Organization for Research and Treatment of Cancer Quality of Life questionnaire (EORTC-QLQ-C30) in patients with pretreated metastatic CRC treated with Napabucasin plus biweekly FOLFIRI versus Napabucasin.
Overall Survival in biomarker positive patients | 43 months
  To assess the effect of Napabucasin plus FOLFIRI versus Napabucasin on the Overall Survival of patients with metastatic colorectal cancer in biomarker positive patients. This biomarker-positive sub-population is defined as those patients with phospho-STAT3/nuclear β-catenin positivity on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) archival tissue.
Progression Free Survival in biomarker positive patients | 43 months
  Defined as the time from randomization to the first objective documentation of disease progression or death due to any cause. This biomarker-positive sub-population is defined as those patients with nuclear β-catenin and/or phospho-STAT3 positivity on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) archival tissue.
Objective Response Rate in biomarker positive patients | 43 months
  Defined as the proportion of patients with a documented complete response or partial response (CR + PR) based on RECIST 1.1. This biomarker-positive sub-population is defined as those patients with nuclear β-catenin and/or phospho-STAT3 positivity on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) archival tissue.Defined as the proportion of patients with a documented complete response or partial response (CR + PR) based on RECIST 1.1. This biomarker-positive sub-population is defined as those patients with nuclear β-catenin and/or phospho-STAT3 positivity on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) archival tissue.
Disease Control Rate in biomarker positive patients | 43 months
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1. This biomarker-positive sub-population is defined as those patients with nuclear β-catenin and/or phospho-STAT3 positivity on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) archival tissue.

CONTACTS AND LOCATIONS:
Locations (37):
- China (37):
  - First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijng Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat - sen University, Guangzhou, Guangdong
  - Forth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The 81 Hospital of the Chinese People's Liberation Army, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Provence Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Liaoning Provincial Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital Qingdao University, Qingdao, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Ren Ji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi' AnJiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang